CLINICAL TRIAL: NCT01747343
Title: Changing the Number of Accidents, Percentage of Appropriate Eliminations, and Number of Self-Initiations Across Toddlers and Preschoolers
Brief Title: Toilet Training Toddlers and Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSCL-17816
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Incontinence; Enuresis
Keywords: Incontinence; Enuresis
MeSH Terms: conditions — Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Underwear/Differential Reinforcement (Experimental): All subjects will wear underwear followed by wearing underwear while receiving differential reinforcement.
  Interventions: Behavioral: Underwear/Differential Reinforcement

INTERVENTIONS:
Behavioral: Underwear/Differential Reinforcement — Participants are going to be placed in underwear. Differential reinforcement will then be implemented.

SUMMARY:
The investigators are interested in determining those procedures that prove to be most efficient and effective in facilitating continence (i.e., "dry pants" or the absence of soiled undergarments), appropriate eliminations (i.e., voids/stools in toilet), and independent requests/initiations to use the toilet. To assess the effectiveness of toilet training methods (procedures), data on toileting skills (in addition to each skill in a given child's curriculum) are collected across the school day (7:30 am-5:45 pm) by the classroom teachers. The primary dependent variables (toileting skills) are continence (i.e., absence of soiled undergarments), appropriate eliminations (i.e., the number of voids/stools made in the toilet), and independent/self requests (i.e., communication by the child with an adult to use the toilet). The toileting procedures are implemented by classroom teachers (undergraduate practicum students) and implementation is monitored by classroom supervisors (graduate teaching assistants). Procedural effectiveness is evaluated on a daily basis by the graduate teaching assistants and on an at-least-weekly basis by faculty supervisors.

DETAILED DESCRIPTION:
First, the effects of the baseline toileting program are assessed. Baseline consists of prompting the child to use the bathroom approximately every 90 min (or more frequently if they independently request to do so). If the investigators observe low levels of continence, appropriate eliminations, and/or independent/self requests, components of the program are systematically altered to increase success. The ultimate goal is for the child to remain continent throughout the day, independently request (or initiate) toilet use, and appropriately eliminate in the toilet once in the bathroom. The following procedural modifications are made if high levels of success are not observed in baseline:

The first modification is to change the child's undergarment type. Specifically, underwear will be used, and it's effects will be evaluated to determine what effect (if any) underwear has on toileting performance.

The second modification is to conduct an individualized preference assessment to identify types of food and leisure items a given child prefers. This is done by having the child select items from an array (items selected based on direct observations of child and parent/teacher report) and allowing him/her access to the chosen item for a brief period of time. This will generate a list of preferred items/activities ranked in order of relative preference. Subsequently, the highest ranked items from the preference assessment will be arranged as reinforcers for continence, appropriate eliminations, and self-initiations. A third modification is to combine the above modifications to determine whether a combination of toilet training procedures enhances toileting performance (as compare to the implementation of individual toilet training procedures). This modification will be conducted while children wear underwear.

ELIGIBILITY:
Inclusion Criteria:

* Individual not yet toilet trained

Exclusion Criteria:

* None

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Greer, Ph.D., Principal Investigator — Doctoral Student (Graduated)
Locations (1):
- Edna A. Hill Child Development Center at the University of Kansas, Lawrence, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four children were recruited from the Edna A. Hill Child Development Center at the University of Kansas from November 2012 until July 2013.
Pre-assignment Details: No children were excluded from the Study.
Period: Baseline
Arm/Group | Underwear/Differential Reinforcement
Started | 4
Completed | 4
Not Completed | 0
Period: Underwear
Arm/Group | Underwear/Differential Reinforcement
Started | 4
Completed | 4
Not Completed | 0
Period: Underwear/Differential Reinforcement
Arm/Group | Underwear/Differential Reinforcement
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Underwear/Differential Reinforcement
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.02 (0.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Number of Accidents Across Children
Time Frame: 2 months minus baseline
Measure: Mean (Standard Deviation); unit: Accidents
Arm/Group | Underwear/Differential Reinforcement
Number analyzed (Participants) | 4
Accidents | -1.3 (1.3)

2. Secondary Outcome: Change in the Mean Percentage of Appropriate Eliminations Across Children
Time Frame: 2 months minus baseline
Measure: Mean (Standard Deviation); unit: Percentage of opportunities
Arm/Group | Underwear/Differential Reinforcement
Number analyzed (Participants) | 4
Percentage of opportunities | 33.4 (41.3)

3. Other Pre Specified Outcome: Change in the Mean Number of Self-initiations to Sit on the Toilet Across Children
Time Frame: 2 months minus baseline
Measure: Mean (Standard Deviation); unit: Self-initiations
Arm/Group | Underwear/Differential Reinforcement
Number analyzed (Participants) | 4
Self-initiations | 2.7 (4.1)

ADVERSE EVENTS:
Arm/Group | Underwear/Differential Reinforcement
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes